CLINICAL TRIAL: NCT00276861
Title: Phase II Study of Oxaliplatin And Fixed Rate Infusion Gemcitabine as Second Line Therapy for Patients With Metastatic Colon Cancer
Brief Title: Gemcitabine and Oxaliplatin as Second-Line Therapy in Treating Patients With Metastatic Colon Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 20030655; SCCC-2003110 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20050993 (Other: Western Institutional Review Board)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; recurrent colon cancer; stage IV colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and oxaliplatin work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with oxaliplatin works as second-line therapy in treating patients with metastatic or recurrent colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete response and partial response rates in patients with recurrent or progressive colon cancer treated with gemcitabine hydrochloride and oxaliplatin.

Secondary

* Determine the overall and failure-free survival of patients treated with the chemotherapy regimen.
* Determine the duration of response (complete or partial) in patients treated with this regimen.
* Determine the percentage of patients who experience a 50% fall of serum carcinoembryonic antigen levels with a baseline elevation of > 5 U/mL after receiving this regimen.
* Evaluate the toxicity associated with the administration of this regimen in these patients.

OUTLINE: This is a non-randomized study.

Patients receive gemcitabine hydrochloride IV over 100 minutes on day 1 and oxaliplatin IV over 2 hours on day 2. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 1 year.

PROJECTED ACCRUAL: A total of 27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the colon

  * Metastatic or recurrent disease
  * Redocumentation of tumor histology or cytology prior to protocol therapy is not required if documented tumor was confirmed prior to initial therapy
* Measurable disease

  * Lesion of ≥ 1 cm in longest diameter that can be repetitively assessed by radiographic measurement or any lesion of ≥ 2 cm in longest diameter that can be repetitively assessed by physical examination
  * Positive bone scans, osteoblastic or osteolytic bone lesions, pleural effusions, and positive bone marrow biopsies are not considered measurable or evaluable lesions
* Metastatic disease to the brain allowed if emergent radiotherapy for symptomatic CNS disease is not required
* Must have received at least one prior chemotherapy regimen (with or without radiotherapy)

  * One of the prior regimens must include irinotecan hydrochloride, fluorouracil, and leucovorin calcium or irinotecan hydrochloride and other fluoropyrimidine
  * Previous therapy with C-225 and/or bevacizumab is allowed
* .

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Granulocyte count ≥1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 2.0 mg/dL
* Bilirubin < 1.5 mg/dL
* SGOT ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious medical or psychiatric illness that would render chemotherapy unsafe
* No concurrent clinically evident malignancy except inactive nonmelanoma skin cancer, low-grade low-stage bladder carcinoma followed off therapy, or lobular neoplasia of the breast
* No clinical AIDS or known positive HIV serology

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* No investigational agent for at least 30 days prior to study entry
* No chemotherapy within the past 3 weeks
* No radiotherapy for palliation within the past 2 weeks prior to study entry
* No prior oxaliplatin or gemcitabine hydrochloride
* No concurrent participation in another clinical trial
* No other concurrent anticancer therapy including chemotherapy, radiotherapy, hormonal therapy, or immunotherapy
* No other concurrent investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-09; Primary Completion 2006-09 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caio Max S. Rocha Lima, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

REFERENCES:
- [Result] Lopes G, Quesada J, Ahn E, Flores A, Ribeiro A, Rocha-Lima CM. Oxaliplatin and fixed-rate infusional gemcitabine in the second-line treatment of patients with metastatic colon cancer: final results of a Phase II trial prematurely closed as a result of poor accrual. Clin Colorectal Cancer. 2007 Sep;6(9):641-5. doi: 10.3816/CCC.2007.n.032. PMID 17945036

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxaliplatin + Gemcitabine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 58.5 [47 to 72]
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Response Rate as Measured by RECIST Criteria
Description: Complete Response (CR) or Partial Response (PR) as defined by RECIST v 1.0 criteria.
Time Frame: 4 - 6 months
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Single Arm
Number analyzed (Participants) | 10
percentage of particpants | 9.9 [5.6 to 15.8]

2. Secondary Outcome: Time to Progression as Measured by the Kaplan Meyer Curve at Completion of Study Treatment
Description: Number of months from time of enrollment to the date of first documented progression or date of death.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Oxaliplatin + Gemcitabine
Number analyzed (Participants) | 10
months | 4.6 [4.2 to 6.1]

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=10)
Neutropenia (Blood and lymphatic system disorders) | 1 — Grade 3/4
Infection (Infections and infestations) | 1 — Grade 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=10)
Anemia (Blood and lymphatic system disorders) | 7 — Grade 1/2
Leukopenia (Blood and lymphatic system disorders) | 4 — grade 1/2
Diarrhea (Gastrointestinal disorders) | 2 — Grade 1/2
Peripheral Neuropathy (Nervous system disorders) | 2 — Grade 1/2
Nausea (Gastrointestinal disorders) | 1 — Grade 1/2
Weight Loss (General disorders) | 1

LIMITATIONS AND CAVEATS:
Protocol closed prematurely due to low accrual. Only 10 of 27 anticipated patients were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No